CLINICAL TRIAL: NCT00456846
Title: An Open-Label, Phase II Study of Weekly ABI-007 as First Line Therapy for Patients With Metastatic Breast Cancer
Brief Title: First Line Therapy for Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA042
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer, ABI-007, Abraxane
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-007 (Experimental): 100 mg/m^2 ABI-007 was administered by intravenous (IV) infusion over 30 minutes weekly for 3 weeks followed by 1 week rest. Therapy continued until disease progression or unacceptable toxicity.
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007 — 100 mg/m^2 ABI-007 weekly for 3 weeks followed by 1 week rest
  Other Names: Nab-paclitaxel; Abraxane

SUMMARY:
The purpose of this study is to determine the toxicity and anti-tumor activity of nab-paclitaxel 100mg/m^2 administered weekly in a 4-week cycle as first line therapy to patients with metastatic breast cancer who received taxanes as part of their adjuvant therapy and patients who did not receive taxanes as part of their adjuvant therapy.

DETAILED DESCRIPTION:
This is an open-label, phase II study to determine the toxicity and antitumor activity of ABI-007 100 mg/m2 administered weekly for 3 weeks followed by a rest week (4-week cycle) as first line therapy to patients with metastatic breast cancer in the following 2 cohorts: Patients who have received a taxane as part of their adjuvant therapy, and patients who did not receive a taxane as part of their adjuvant therapy. Patients will be assessed for antitumor response every 8 weeks.

The last subject received study treatment 11DEC2012. The study was terminated on 31 May 2013 via a notification letter to all investigators on 14 May 2013.

ELIGIBILITY:
Inclusion Criteria:

* Females with pathologically confirmed adenocarcinoma of the breast.
* No prior chemotherapy for metastatic breast cancer
* At least 12 months between completion of adjuvant chemotherapy and the diagnosis of metastatic disease
* Stage IV disease
* Measurable disease (must be equal or greater to 2.0 cm using conventional Computed Tomography (CT) or equal or greater to 1.0 cm using spiral CT except for pulmonary lesions that are well documented on conventional CT scan which must be equal or greater than 1.0 cm)
* At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal or there must be radiologic or clinical exam proof of progressive disease within the radiation portal
* At least 4 weeks since major surgery, with full recovery
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age equal or greater to 18
* Patients has the following blood counts at Baseline:
* Absolute Neutrophil Count (ANC) equal or greater to 1.5 x 10^9 cells/L
* Platelets equal or greater to 100 x 10^9 cells/L
* Hemoglobin (Hgb) equal or greater to 90 grams/L
* Patients has the following blood chemistry levels at Baseline:
* Aspartate aminotransferase (AST) Serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT) serum glutamic:pyruvic transaminase (SGPT)less than or equal to 2.5x upper limit of normal range (ULN);
* total bilirubin normal (unless bilirubin elevation is due to Gilbert's (Disease);
* alkaline phosphatase less than or equal 2.5x ULN (unless bone metastasis is present in the absence of liver metastasis);
* Creatinine less than or equal to 1.5mg/dL
* Current sensory neuropathy Grade 0 or 1 by Breast Cancer Index (BCI) Common Toxicity Criteria Adverse Events (CTCAE)
* If female of childbearing potential, pregnancy test is negative (within 72 hours of the first dose of study drug).
* If fertile, the patient agrees to use an effective method of contraception to avoid pregnancy for the duration of the study
* Patient is able to supply unstained slides or 1 tumor block of her primary breast tumor or a biopsy of a current site of metastasis for Secreted protein acidic and rich in cysteine (SPARC) analysis
* Informed consent has been obtained

Exclusion Criteria:

* Concurrent immunotherapy or hormonal therapy (other than Herceptin) for breast cancer
* Parenchymal brain metastases, unless documented to be clinically and radiographically stable for at least 6 months after treatment
* Serious intercurrent medical or psychiatric illness, including serious active infection
* History of class II-IV congestive heart failure
* History of other malignancy within the last 5 years which could affect the diagnoses or assessment of breast cancer, with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Patients who have received an investigational drug within the previous 3 weeks
* Patient is currently enrolled in a different clinical study in which investigational procedures are performed or investigational therapies are administered. Also a patient may not enroll in such clinical trials while participating in this study.
* Pregnant or nursing women
* Patients with prior hypersensitivity to Taxol or Taxotere

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2012-12-11 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Smiljanik, MD, Principal Investigator — Lions Gate Hospital; Kara Laing, MD, Principal Investigator — Dr. H. Bliss Murphy Cancer Center; Wendy Lam, MD, Principal Investigator — BC Cancer Agency-Burnaby; Maureen Trudeau, MD, Principal Investigator — Toronto Sunnybrook Cancer Centre; Vanessa Bernstein, MD, Principal Investigator — B.C.C.A. Vancouver Island Center; Jawaid Younus, MD, Principal Investigator — London Regional Cancer Centre; Lawrence Panasci, MD, Principal Investigator — McGill University; Guy Cantin, MD, Principal Investigator — CHA: Saint Sacrement Hospital; Nicolas Raymond, MD, Principal Investigator — Hospital de la Cite-de-la Sante-de-Laval; Robert El-Maraghi, MD, Principal Investigator — The Royal Victoria Hospital; Christine Brezden-Masley, MD, Principal Investigator — Unity Health Toronto; Andre Robidoux, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal-Hotel-Dieu; Martin Blackstein, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Caroline Hamm, MD, Principal Investigator — Windsor Regional Cancer Center
Locations (14):
- Canada (14):
  - BC Cancer Agency-Burnaby, Burnaby, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - B.C.C.A Vancouver Island Center, Victoria, British Columbia
  - Dr. H. Bliss Murphy Cancer Center, St. John's, Newfoundland and Labrador
  - The Royal Victoria Hospital, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Synnybrook Cancer Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Hospital de la Cite-de-la Sante-de-Laval, Laval, Quebec
  - Centre Hospitalier de l'Universite de Montreal-Hotel-Dieu, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - CHA: Saint Sacrement Hospital, Québec

REFERENCES:
- [Background] Brezden B, et al. An open-label, phase II study of weekly nab-paclitaxel as first-line therapy for patients (pts) with metastatic breast cancer (MBC): Safety update. Presented at 2010 ASCO Annual Meeting, June 4-8, 2010, Chicago, IL. Abstract No 1127 C.

RESULTS

PARTICIPANT FLOW:
Groups:
- Abraxane (Prior Taxane Therapy): Participants who had received a taxane as part of their adjuvant therapy received Abraxane (ABI-007) at 100 mg/m^2 given intravenously (IV) over 30 minutes weekly for 3 weeks followed by 1 week rest. Therapy continued until disease progression or unacceptable toxicity.
- Abraxane (No Prior Taxane Therapy): Participants who had not received a taxane as part of their adjuvant therapy received Abraxane (ABI-007) at 100 mg/m^2 given intravenously (IV) over 30 minutes weekly for 3 weeks followed by 1 week rest. Therapy continued until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Started | 47 | 76
Completed | 31 (Treatment considered completed upon disease progression) | 48 (Treatment considered completed upon disease progression)
Not Completed | 16 | 28
Not completed — Adverse Event | 2 | 15
Not completed — Physician Decision | 11 | 6
Not completed — Protocol Deviation | 2 | 0
Not completed — Participant Discretion | 1 | 5
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated Population
Groups:
- Abraxane (Prior Taxane Therapy): Participants who had received a taxane as part of their adjuvant therapy received Abraxane (ABI-007) at 100 mg/m^2 given intravenously (IV) over 30 minutes weekly for 3 weeks followed by 1 week rest
- Abraxane (No Prior Taxane Therapy): Participants who had not received a taxane as part of their adjuvant therapy received Abraxane (ABI-007) at 100 mg/m^2 given intravenously (IV) over 30 minutes weekly for 3 weeks followed by 1 week rest
- Total: Total of all reporting groups
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy) | Total
Number analyzed (Participants) | 47 | 76 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.78) | 58.3 (10.88) | 57.2 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 76 | 123
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 5 | 5
  Black, of African Heritage | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White, Non-Hispanic/Non Latino | 41 | 60 | 101
  White, Hispanic or Latino | 0 | 5 | 5
  Other-Unspecified | 3 | 3 | 6
Menopausal Status [Number; unit: participants]
  Premenopausal | 12 | 12 | 24
  Postmenopausal | 35 | 64 | 99
Stage at Primary Diagnosis [Number; unit: participants] — Invasive breast cancer stages:
  Stage I-cancer cells are breaking through to or invading normal surrounding breast tissue.
  Stage IIa-breast tumor about 2cm and involvement of ancillary lymph nodes. Stage IIb-a larger tumor than earlier phases. Stage IIIa-axillary lymph nodes clumping together. Stage IIIb-spread further to the skin, breast bone or chest wall. Stage IIIc-expanded involvement of lymph nodes. Stage IV-cancer that has spread beyond the breast and nearby lymph nodes to other organs of the body.
  participants
    Stage I | 4 | 12 | 16
    Stage IIa | 7 | 12 | 19
    Stage IIb | 14 | 13 | 27
    Stage IIIa | 11 | 8 | 19
    Stage IIIb | 6 | 4 | 10
    Stage IIIc | 5 | 5 | 10
    Stage IV | 0 | 19 | 19
    Unknown | 0 | 3 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used to assess the progress of disease in a patient, how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  participants
    0 (fully active) | 21 | 38 | 59
    1 (restrictive but ambulatory) | 22 | 30 | 52
    2 (ambulatory but unable to work) | 4 | 8 | 12
    3 (limited self-care) + 4 (completely disabled) | 0 | 0 | 0
Physician Assessment of Peripheral Neuropathy] [2] [Number; unit: participants] — The physician assessed sensory neuropathy using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) of "Neurology -- Neuropathy - Sensory". The scale is 0 = normal, 1 = asymptomatic; loss of deep tendon reflexes or paresthesia (including tingling) but not interfering with function, 2 = sensory alteration or paresthesia (including tingling), interfering with activities of daily living (ADL); 3 = Sensory alteration or parasthesia interfering with ADLs; 4 = disabling
  participants
    Grade 0 | 37 | 69 | 106
    Grade 1 | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Confirmed Complete or Partial Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 Based on Investigator and Independent Reviewers
Description: Overall response rate (ORR) is complete response (CR) + partial response (PR). Complete response (CR): The disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation. All sites must be assessed, including non-measurable sites, such as effusions, or markers. Disappearance of all non-target lesions. The normalization of tumor marker level confirmed at least 4 weeks after initial documentation. Partial response (PR): At least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing. As well as persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits
Time Frame: Every 8 weeks from study start until disease progression; Up to 61 months
Population: Treated Population: The Treated population consisted of all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
percentage of participants
  Investigator Assessment | 30 [16.7 to 42.9] | 28 [17.6 to 37.7]
  Independent Reviewer Assessment | 32 [18.6 to 45.2] | 32 [21.1 to 42.0]

2. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control was defined as stable disease (SD) for ≥ 16 weeks or complete response (CR) or partial response (PR). Response was evaluated by the Investigator and by an independent reviewer using Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.0. See Outcome #1 for definitions of CR and PR. RECIST defines SD for target lesions as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: Every 8 weeks from study start until disease progression; Up to 61 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
percentage of participants
  Investigator Assessment | 51 [36.8 to 65.4] | 57 [45.4 to 67.7]
  Independent Reviewer Assessment | 55 [41.1 to 69.5] | 57 [45.4 to 67.7]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose of study drug to the start of progression or patient death (any cause), whichever occurred first. Participants who did not have progression or did not die were censored at the last known time the participant was progression free. Participants who initiated other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
Time Frame: Study start until disease progression, death, or up to data cut off of 31 May 2013; up to 61 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
months
  Investigator Assessment | 6.0 [3.5 to 8.8] | 6.7 [5.3 to 7.3]
  Independent Reviewer Assessment | 5.3 [3.3 to 7.3] | 5.3 [3.5 to 6.6]

4. Secondary Outcome: Duration of Response Based on Independent Reviewer Assessment
Description: Duration of response was defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or patient death from any cause, whichever occurred first. Participants who did not have progression or had not died were censored at the last known time the participant was progression free. Participants who had initiated other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated. CR and PR were defined in outcome #1. Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion. Response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Initial response until disease progression; or until data cut off 31 May 2013; up to 61 months
Population: Treated Population: The Treated population with a confirmed complete response or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 15 | 24
months | 10.9 [7.3 to 18.9] | 9.2 [7.4 to 14.2]

5. Secondary Outcome: Duration of Response Based on Investigator Assessment
Description: Duration of response was defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or patient death from any cause, whichever occurred first. Participants who did not have progression or had not died were censored at the last known time the participant was progression free. Participants who had initiated other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated. Complete response (CR) and partial response (PR) were defined in outcome #1. Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion. Response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Initial response until disease progression; or until data cut off 31 May 2013; up to 61 months
Population: Treated Population: The Treated population consisted of all enrolled participants that received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 14 | 21
months | 10.5 [8.8 to 25.4] | 10.8 [8.7 to 22.4]

6. Secondary Outcome: Patient Survival
Description: Participant survival was the time from the first dose of study drug to participant death from any cause. Participants who did not die were censored at the last known time the participant was alive.
Time Frame: Study start until death, or until data cut-off 31 May 2013; up to 61 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
months | 20.9 [14.3 to 28.0] | 20.0 [13.8 to 28.6]

7. Secondary Outcome: Number of Participants Experiencing Dose Reductions, Interruptions, or Dose Delays of Study Drug
Description: The number of participants with dose reductions, dose interruptions and dose delays that occurred during the treatment period. Dose reductions, interruptions and delays are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
Time Frame: Day 1 of study drug to Day 940; data cut off 31 May 2013
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
participants
  Patients with at Least One Dose Reduction | 11 | 19
  Patients with at Least One Dose Interruption | 3 | 2
  Patients with at Least One Dose Delay/Not Given | 20 | 39

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Count of study participants who had at least one treatment-emergent adverse event (TEAE) defined as any adverse event that began or worsened in grade after the start of study drug through 30 days after the last dose of study drug. The National Cancer Institute (NCI)'s Common Terminology Criteria for AEs (CTCAE) was used to grade AE severity: severity grade 3= severe and undesirable AE. Severity grade 4= life-threatening or disabling AE. Severity grade 5 = death.
Time Frame: Day 1 to Day 940
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Number analyzed (Participants) | 47 | 76
participants
  ≥1 Adverse Event (AE) | 46 | 75
  ≥1 Treatment related Adverse Event | 41 | 74
  ≥ 1 Serious Adverse Event | 5 | 14
  Treatment related Serious Adverse Event | 2 | 7
  ≥1 One Grade 3/4 Adverse Event | 25 | 36
  ≥1 One Grade 3 or Higher Adverse Event | 25 | 36
  ≥1 AE leading to treatment discontinuation | 2 | 16
  ≥1 AE leading to death | 0 | 2
  ≥1 AE leading to dose reduction of study drug | 11 | 18
  ≥1 AE leading to dose interruption of study drug | 2 | 0
  ≥1 AE leading to dose delay of study drug | 15 | 29

ADVERSE EVENTS:
Time Frame: Any Adverse Event (AE) that started after initial study drug administration through the end of the study or 30 days after the last treatment, whichever was later, were followed until the AE had resolved or stabilized. Upt to 61 months.
Arm/Group | Abraxane (Prior Taxane Therapy) | Abraxane (No Prior Taxane Therapy)
Serious Adverse Events (participants affected / at risk) | 5/47 | 14/76
Other Adverse Events (participants affected / at risk) | 46/47 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane (Prior Taxane Therapy) (N=47) | Abraxane (No Prior Taxane Therapy) (N=76)
Pneumonia (Infections and infestations) | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane (Prior Taxane Therapy) (N=47) | Abraxane (No Prior Taxane Therapy) (N=76)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Dry eye (Eye disorders) | 1 | 5
Lacrimation increased (Eye disorders) | 5 | 14
Vision blurred (Eye disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 12
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 15 | 15
Diarrhoea (Gastrointestinal disorders) | 15 | 37
Dry mouth (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 11 | 9
Dysphagia (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 24 | 47
Stomatitis (Gastrointestinal disorders) | 6 | 18
Vomiting (Gastrointestinal disorders) | 13 | 22
Asthenia (General disorders) | 5 | 6
Chills (General disorders) | 6 | 5
Fatigue (General disorders) | 33 | 55
Influenza like illness (General disorders) | 1 | 5
Mucosal inflammation (General disorders) | 1 | 4
Non-cardiac chest pain (General disorders) | 3 | 4
Oedema (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 13 | 22
Pain (General disorders) | 4 | 3
Performance status decreased (General disorders) | 2 | 6
Pyrexia (General disorders) | 8 | 17
Cellulitis (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Urinary tract infection (Infections and infestations) | 6 | 8
Fall (Injury, poisoning and procedural complications) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 5
Haemoglobin decreased (Investigations) | 4 | 9
Neutrophil count decreased (Investigations) | 0 | 4
Weight decreased (Investigations) | 6 | 6
Weight increased (Investigations) | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 16 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 15
Dizziness (Nervous system disorders) | 10 | 17
Dysgeusia (Nervous system disorders) | 10 | 19
Headache (Nervous system disorders) | 17 | 20
Hypoaesthesia (Nervous system disorders) | 5 | 4
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 44
Somnolence (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 3 | 10
Depression (Nervous system disorders) | 5 | 5
Insomnia (Nervous system disorders) | 6 | 15
Mood altered (Nervous system disorders) | 1 | 4
Urinary incontinence (Renal and urinary disorders) | 0 | 4
Breast pain (Reproductive system and breast disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 61
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 12 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 14
Hot flush (Vascular disorders) | 4 | 11
Hypertension (Vascular disorders) | 1 | 4
Lymphoedema (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to their submission; Celgene shall complete its review within 60 days after receipt. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of patentable material.